CLINICAL TRIAL: NCT05857488
Title: Feasibility, Safety and Utility of Endomicroscopy to Study the Intestines of Unsedated Infants at University of Virginia (UVa)
Brief Title: Feasibility, Safety and Utility of Endomicroscopy to Study the Intestines of Unsedated Infants at UVa
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A shift occurred in the focus of the research, following the emergence of new scientific knowledge regarding the disease. Hence, study was terminated early and withdrawn by the investigator and no further subjects were enrolled.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2021P003264
Record Dates: First submitted 2023-03-09; First posted 2023-05-12 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: OCT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Trans Nasal Endomicroscopy Imaging (Experimental): The subject will have the transnasal introduction tube inserted, and OCT images will be acquired using the OCT compact imaging system. The subject may also undergo a microbiome brushing and/or intestinal potential difference measurement procedure during the study visit.
  Interventions: Device: Transnasal introduction tube

INTERVENTIONS:
Device: Transnasal introduction tube — Imaging of the GI tract using the transnasal introduction tube and system. Optional gut microbiome sample collection using the microbiome brush and/or intestinal potential difference measurement using the intestinal potential difference probe.
  Other Names: Microbiome brush; Intestinal potential difference probe

SUMMARY:
The purpose of this study is to demonstrate the feasibility of using the transnasal endomicroscopy (TNE) platform, using intestinal potential difference (IPD) and microbiome brush to evaluate the intestine of unsedated infants.

DETAILED DESCRIPTION:
A total of fifteen (15) subjects, infants 6 months of age to 48 months of age will be enrolled in this study.

While the subject is awake and unseated, a catheter with optical coherence tomography (OCT) imaging technology will be introduced transnasally. Images will be acquired while the tube is moved through the subject's GI tract. After imaging is complete, accessory device(s) may be threaded through the catheter to collect samples of the gut microbiome and/or measure intestinal potential difference.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 48 month old infants that can follow fasting requirements

Exclusion Criteria:

* Any infant under 6kg of weight since this is the minimum weight for 6.5 F nasogastric (NG) tube
* Any infant whose nasal passage cannot reasonably accommodate a 6.5 French nasoduodenal catheter.
* Any infants with absolute or relative contraindications to transnasal tubes:

  1. severe midface trauma and recent nasal, throat, or esophageal surgery.
  2. Esophageal varices, esophageal stricture, and alkaline ingestion
  3. Congenital anatomical defects affecting the gastrointestinal tract, most specifically cleft lip and/or cleft palate.
* Any infant with absolute or relative contraindication to a duodenal biopsy:

  1. post bone marrow transplant
  2. coagulation abnormalities

Ages: 6 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- University of Virginia Children's Hospital, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trans Nasal Endomicroscopy Imaging
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Trans Nasal Endomicroscopy Imaging
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 27 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Ability to Acquire Intestinal Images in an Unsedated Infant
Description: Can the technology successfully collect images of the small intestine in an unseated infant?
Time Frame: Approximate 90 minute study visit
Population: Procedure was terminated early due to loss of the imaging signal, therefore no OCT images of the small intestines were acquired for this subject, thus this participant could not be assessed for this outcome measure.
Arm/Group | Trans Nasal Endomicroscopy Imaging
Number analyzed (Participants) | 0

2. Primary Outcome: Ability for Unsedated Infant Subjects to Tolerate the Device
Description: Can the unsedated infant subjects tolerate the administration of the device with minimal discomfort?
Time Frame: Approximate 90 minute study visit
Population: The procedure was tolerated by the study participant during insertion, imaging of the stomach and removal of the TNIT but the procedure was terminated early due to loss of imaging signal while in the stomach, with no clinical or safety impact on the study participant. Tolerability could not be assessed for some portions of the study procedure including transit to the small intestine, IPD measurements and microbiome brush sample collection.
Measure: Count of Participants; unit: Participants
Arm/Group | Trans Nasal Endomicroscopy Imaging
Number analyzed (Participants) | 1
Participants | 1

3. Primary Outcome: Ability to Visualize Features of the Small Intestine in Unsedated Infants.
Description: Can the technology successfully visualize features of the small intestine (villi etc) on OCT in unsedated infants?
Time Frame: Approximate 90 minute study visit
Population: OCT images were acquired through the TNIT from the esophagus and stomach but the procedure was terminated early due to loss of imaging signal while in the stomach, with no clinical or safety impact on the study participant. Features of the small intestine (villi etc) could not be assessed.
Arm/Group | Trans Nasal Endomicroscopy Imaging
Number analyzed (Participants) | 0

4. Primary Outcome: Ability to Acquire Microbiome Brush and Intestinal Potential Difference Samples
Description: Can the technology successfully collect microbiome brush and/or intestinal potential differences samples?
Time Frame: Approximate 90 minute study visit
Population: The procedure was terminated early and target samples were not collected in the enrolled subject. Subsequently, a shift occurred in the focus of the research, following the emergence of new scientific knowledge regarding the disease. Hence, study was terminated early and withdrawn by the investigator and no further subjects were enrolled.
Arm/Group | Trans Nasal Endomicroscopy Imaging
Number analyzed (Participants) | 0

5. Secondary Outcome: Amount and Composition of Microbial Samples Acquired Via Microbiome Brush Sampling in Unsedated Infants
Description: Measurements including DNA load and microbial composition will be collected.
Time Frame: Approximate 90 minute study visit
Population: as for outcome 4
Arm/Group | Trans Nasal Endomicroscopy Imaging
Number analyzed (Participants) | 0

6. Secondary Outcome: Ability to Collect Intestinal Potential Difference Measurements in Various Locations in the Gastrointestinal Tract of Unsedated Infants
Description: Intestinal potential difference measurements will be collected at various locations to determine the feasibility of measuring IPD in unsedated infants
Time Frame: Approximate 90 minute study visit
Population: The procedure was terminated early prior to the TNIT entering the small intestine due to loss of imaging signal while in the stomach, with no clinical or safety impact on the study participant and IPD measurements were not collected.
Arm/Group | Trans Nasal Endomicroscopy Imaging
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The duration of the imaging procedure (approximate 90 minute study visit) and post visit follow up phone call, the following day.
Description: No adverse event has been reported
Arm/Group | Trans Nasal Endomicroscopy Imaging
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT05857488/Prot_SAP_000.pdf